CLINICAL TRIAL: NCT00769288
Title: A Phase I Study of Intravenously Administered FAU (1-(2'-Deoxy-2'-Fluoro-B-D-arabinofuranosyl) Uracil, NSC#678515) in Patients With Advanced Solid Tumors
Brief Title: FAU in Treating Patients With Advanced Solid Tumors or Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00248; NCI-2009-00248 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000615651; WSU#2007-005; WSU-2007-005 (Other: Wayne State University); 7916 (Other: CTEP); P30CA022453 (NIH); U01CA062487 (NIH)
Record Dates: First submitted 2008-10-08; First posted 2008-10-09 (Estimated); Last update posted 2014-01-07 (Estimated); Status verified 2014-01

CONDITIONS: Adult Grade III Lymphomatoid Granulomatosis; Adult Nasal Type Extranodal NK/T-cell Lymphoma; Anaplastic Large Cell Lymphoma; Angioimmunoblastic T-cell Lymphoma; Cutaneous B-cell Non-Hodgkin Lymphoma; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Nodal Marginal Zone B-cell Lymphoma; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Adult Grade III Lymphomatoid Granulomatosis; Recurrent Adult Hodgkin Lymphoma; Recurrent Adult Immunoblastic Large Cell Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Adult T-cell Leukemia/Lymphoma; Recurrent Cutaneous T-cell Non-Hodgkin Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Mycosis Fungoides/Sezary Syndrome; Recurrent Small Lymphocytic Lymphoma; Small Intestine Lymphoma; Splenic Marginal Zone Lymphoma; Stage III Adult Burkitt Lymphoma; Stage III Adult Diffuse Large Cell Lymphoma; Stage III Adult Diffuse Mixed Cell Lymphoma; Stage III Adult Diffuse Small Cleaved Cell Lymphoma; Stage III Adult Hodgkin Lymphoma; Stage III Adult Immunoblastic Large Cell Lymphoma; Stage III Adult Lymphoblastic Lymphoma; Stage III Adult T-cell Leukemia/Lymphoma; Stage III Cutaneous T-cell Non-Hodgkin Lymphoma; Stage III Grade 1 Follicular Lymphoma; Stage III Grade 2 Follicular Lymphoma; Stage III Grade 3 Follicular Lymphoma; Stage III Mantle Cell Lymphoma; Stage III Marginal Zone Lymphoma; Stage III Mycosis Fungoides/Sezary Syndrome; Stage III Small Lymphocytic Lymphoma; Stage IV Adult Burkitt Lymphoma; Stage IV Adult Diffuse Large Cell Lymphoma; Stage IV Adult Diffuse Mixed Cell Lymphoma; Stage IV Adult Diffuse Small Cleaved Cell Lymphoma; Stage IV Adult Hodgkin Lymphoma; Stage IV Adult Immunoblastic Large Cell Lymphoma; Stage IV Adult Lymphoblastic Lymphoma; Stage IV Adult T-cell Leukemia/Lymphoma; Stage IV Cutaneous T-cell Non-Hodgkin Lymphoma; Stage IV Grade 1 Follicular Lymphoma; Stage IV Grade 2 Follicular Lymphoma; Stage IV Grade 3 Follicular Lymphoma; Stage IV Mantle Cell Lymphoma; Stage IV Marginal Zone Lymphoma; Stage IV Mycosis Fungoides/Sezary Syndrome; Stage IV Small Lymphocytic Lymphoma; Unspecified Adult Solid Tumor, Protocol Specific; Waldenström Macroglobulinemia
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Lymphoma, B-Cell, Marginal Zone; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Leukemia, Lymphocytic, Chronic, B-Cell; Waldenstrom Macroglobulinemia | interventions — 2'-fluoro-5-ethylarabinosyluracil; Magnetic Resonance Spectroscopy; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole; Pharmacogenomic Testing

ARMS (1):
- I (Experimental): Patients will receive a 1-hour infusion of FAU on days 1-5.
  Interventions: Drug: 2'-F-ara-deoxyuridine; Other: positron emission tomography; Other: laboratory biomarker analysis; Other: pharmacological study; Other: pharmacogenomic studies

INTERVENTIONS:
Drug: 2'-F-ara-deoxyuridine — Given IV
  Other Names: FAU
Other: positron emission tomography — Correlative studies
  Other Names: FDG-PET; PET; PET scan; tomography, emission computed
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: pharmacogenomic studies — Correlative studies
  Other Names: Pharmacogenomic Study

SUMMARY:
Drugs used in chemotherapy, such as FAU, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. This phase I trial is studying the side effects and best dose of FAU in treating patients with advanced solid tumors or lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety and tolerability of FAU in patients with advanced solid tumors or lymphoma.

II. To determine the dose-limiting toxicity and maximum tolerated dose (MTD) of FAU in these patients.

SECONDARY OBJECTIVES:

I. To observe the clinical response in patients treated with FAU. II. To characterize the pharmacokinetics of FAU in these patients. III. To explore whether an association exists between pre-treatment 18F-FAU PET standardized uptake value levels and time to tumor progression after treatment with unlabeled FAU.

IV. To estimate the protein levels of thymidylate synthase (TS) in archival tumor tissue samples and to compare them with thymidine kinase (TK) and TS protein levels and TK and TS mRNA levels in fresh tumor tissue samples from patients treated at the MTD.

V. To explore the relationship between genetic polymorphisms of TS and tumor 18F-FAU uptake.

OUTLINE: This is a multicenter study.

Patients receive FAU IV over 1 hour on days 1-5. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Measurable disease by CT scan and/or MRI
* Archival tumor tissue sample available for correlative pharmacodynamic and pharmacogenomic studies
* Accessible tumor tissue available (for patients enrolled in the expanded maximum tolerated dose [MTD] cohort)
* No known active brain metastases but previously treated brain metastases allowed
* ECOG performance status (PS) 0-1 OR Karnofsky PS 70-100%
* AST and ALT =< 2.5 times upper limit of normal (ULN) (=< 5 times ULN if liver metastases are present)
* Alkaline phosphatase =< 2.0 times ULN (=< 5 times ULN if bone or liver metastases are present)
* Bilirubin normal
* Creatinine normal or creatinine clearance >= 60 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Willing to undergo tumor biopsies for correlative pharmacodynamic studies (for patients enrolled in the expanded MTD cohort)
* Able to lie still for PET scan
* Weight =< 300 lbs
* No uncontrolled illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness/social situation that would preclude compliance with study requirements
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to FAU
* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas, mitomycin C, or bleomycin), immunotherapy, or experimental therapy and recovered
* More than 4 weeks since prior radiotherapy to > 5% of total marrow volume
* No prior radiotherapy to >= 50% of total marrow volume
* More than 3 weeks since prior radiotherapy to =< 5% of total marrow volume
* No other concurrent investigational agents
* ANC >= 1,500/mm^3
* Platelet count >= 100,000/mm^3
* Life expectancy > 12 weeks
* Histologically or cytologically confirmed malignant solid tumor for which standard curative or palliative measures do not exist or are no longer effective
* Solid hematologic malignancies (e.g., Hodgkin or non-Hodgkin lymphoma) allowed provided bone marrow biopsy has been performed within the past 6 weeks
* Metastatic or unresectable disease
* No other concurrent anticancer therapy (e.g., cytotoxic therapy, biologic therapy, radiotherapy, or hormonal therapy)
* Concurrent hormone replacement therapy allowed
* Concurrent megestrol acetate or bisphosphonates allowed provided they were started 1 month prior to study enrollment
* Concurrent luteinizing hormone-releasing hormone agonists to maintain castrate levels of testosterone allowed for patients with prostate cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-07; Primary Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose, defined as the dose at which no more than 1/6 patients develops dose-limiting toxicity, graded by NCI CTCAE version 4.0 | Up to 28 days

SECONDARY OUTCOMES:
Clinical response to FAU, evaluated using the new international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) Committee | Up to 30 days
  Response will be described by point estimates and exact confidence intervals.
Pharmacokinetics of FAU, including Cmax, Tmax, AUC 0-last, AUC 0-infinity, CL, t1/2, and Vss | Days 1 and 22 of course 1 at pre-treatment; at the end of infusion; and following the end of infusion at 15 and 30 minutes and 1, 2, 4, 8, and 24 hours
  All pharmacokinetic parameters will be summarized with standard descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia LoRusso, Principal Investigator — Wayne State University
Locations (1):
- Wayne State University, Detroit, Michigan, United States